CLINICAL TRIAL: NCT03986892
Title: Functional Aging in Health and Heart Failure: The COmPLETE Study
Brief Title: The COmPLETE Study
Acronym: COmPLETE
Status: Completed | Type: Observational
Sponsor: Arno Schmidt-Trucksäss (Other)
Responsible Party: Sponsor-Investigator, Arno Schmidt-Trucksäss, Prof. Dr. med., University of Basel
Organization: University of Basel (Other)
Other Study IDs: 182815
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Aging; Heart Failure
Keywords: fitness; exercise; vascular function
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COmPLETE-Health: No intervention
  Interventions: Behavioral: Physical Activity
- COmPLETE-Heart: No intervention
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Physical Activity

SUMMARY:
The project is designed as a large scale, cross-sectional study. This research seeks to identify physical fitness and cardiovascular parameters that best resemble underlying cardiovascular risk with age. Further, it will examine which physical fitness markers are impaired most in heart failure.

DETAILED DESCRIPTION:
Cardiovascular (CV) diseases including heart failure are the leading causes of morbidity, with age being the primary risk factor. The combination of age-related organic functional impairment and reduced physical fitness can drastically impact an individual's healthspan. One's lifespan can potentially be prolonged by the preservation or improvement of physical fitness. However, it remains unclear as to which biomarkers are most suitable for distinguishing between healthy aging and the impaired organ function associated with heart failure. Therefore, a comprehensive assessment of the components of physical fitness and CV function will be performed to identify the most important factors contributing to aging in relation to both health and disease.

This cross-sectional investigation will consist of two parts: the COmPLETE-Health (C-Health) and COmPLETE-Heart (C-Heart) studies. C-Health will examine the aging trajectories of physical fitness components and CV properties in a healthy population sample aged between 20 and 100 years (n = 490). Separately, C-Heart will assess the same markers in patients at different stages of chronic heart failure (n = 80). The primary outcome to determine the difference between C-Health and C-Heart will be cardiorespiratory fitness as measured by cardiopulmonary exercise testing on a bicycle ergometer. Secondary outcomes will include walking speed, balance, isometric strength, peak power, and handgrip strength. Physical activity as a behavioural component will be assessed objectively via accelerometry. Further, CV assessments will include pulse wave velocity; retinal, arterial, and venous diameters; brachial and retinal arterial endothelial function; carotid intima-media thickness; and systolic and diastolic function. The health distances for C-Health and C-Heart will be calculated using the methodology based on statistical (Mahalanobis) distance applied to measurements of quantitative biomarkers.

This research seeks to identify physical fitness and CV biomarkers that best resemble underlying CV risk with age. Further, it will examine which physical fitness markers are impaired most in heart failure. The presented integrative approach could define new recommendations for diagnostic guidance in aging. Ultimately, this study is expected to offer a better understanding of which functional characteristics should be specifically targeted in primary and secondary prevention to achieve an optimal healthspan.

ELIGIBILITY:
Inclusion Criteria

C-Health:

• Healthy men and women aged 20-100 years

* Body mass index < 30 kg/m2
* Nonsmoker

C-Heart:

* Stable CHF (treated patient with symptoms and signs that have remained generally unchanged for at least one month) characterized according to the European Society of Cardiology guidelines for the diagnosis and treatment of acute and chronic heart failure [82], as follows:

  1. HFrEF (LVEF < 40%)
  2. HFmHF (LVEF 40-49%)
  3. HFpEF (LVEF ≥ 50%) and NT-proBNP > 125 pg/mL and structural or functional changes in echocardiography in no. 2 or 3.

     Exclusion criteria

     C-Health:
* Age younger than 20 years; manifest exercise limiting chronic disease (e.g., myocardial infarction; stroke; heart failure; lower-extremity artery disease; cancer with general symptoms; diabetes; clinically apparent renal failure; severe liver disease; chronic bronchitis GOLD stages II to IV; osteoporosis), women with known pregnancy or breastfeeding; drug or alcohol abuse; hypertonic blood pressure of less than 160/100 mmHg; compromising orthopaedic problems; Alzheimer's disease or any other form of dementia; inability to follow the procedures of the study (e.g., due to language problems, psychological disorders, dementia of the participant); diseases regarded as an absolute contraindication for maximal exertion; and current or past smoking status.

C-Heart:

• Age younger than 20 years; women with known pregnancy or breastfeeding; drug or alcohol abuse; inability to follow the study procedures (e.g., due to language problems, psychological disorders, etc.); unstable angina pectoris; uncontrolled brady- or tachyarrythmia; paroxysmal atrial fibrillation; severe uncorrected valvular disease; acute myocardial infarction or coronary syndrome; transient ischemic attack or stroke occurring less than three months prior; clinically significant concomitant disease states (e.g. uncontrolled hypertonic blood pressure); clinical evidence of current malignancy with exception of basal cell or squamous cell carcinoma of the skin and/or cervical intraepithelial neoplasia; currently receiving systemic chemotherapy and/or radiotherapy; significant musculoskeletal disease other than that associated with heart failure limiting exercise tolerance; active infection; immunosuppressive medical therapy; life-expectancy of less than six months; and prevalence of a disease regarded as an absolute contraindication for maximal exertion.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In C-Health, recruitment will be performed until a total number of 490 participants with a valid cardiopulmonary exercise test (CPET) as our primary outcome are included. All participants will be recruited in the area of Basel, including 35 males and 35 females per age category (i.e., 20-29, 30-39, 40-49, 50-59, 60-69, 70-79, and 80+ years of age).
  C-Heart will include 80 heart failure patients characterized according to criteria named below.
  Stable CHF (treated patient with symptoms and signs that have remained generally unchanged for at least one month) characterized according to the European Society of Cardiology guidelines for the diagnosis and treatment of acute and chronic heart failure [82], as follows:
  1. HFrEF (LVEF < 40%)
  2. HFmHF (LVEF 40-49%)
  3. HFpEF (LVEF ≥ 50%) and NT-proBNP > 125 pg/mL and structural or functional changes in echocardiography in no. 2 or 3.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratroy Fitness | 3 hours after inclusion in study
  Maximal Oxygen uptake measured by cardiopulmonary exercise testing (VO2peak) in L/min
Ventilatory Efficiency | 3 hours after inclusion in study
  VE/VCO2 measured by cardiopulmonary exercise testing ((L/min)/(L/min))
Oxygen Uptake Efficiency | 3 hours after inclusion in study
  The Oxygen Uptake Efficiency Slope is defined as the regression slope 'a' in V̇O2 = a × log VE +b measured by cardiopulmonary exercise testing.
Gait speed | 1.5 hours after inclusion in study
  Gait speed measured by an inertial sensor system in m/s.
Standing balance | 2.5 hours after inclusion in study
  The cumulative sway path (cm) serves as a measure of postural control.
Hand grip strength | 2.5 hours after inclusion in study
  Measured by a handheld dynamometer. Maximal achieved grip strength (kg) is recorded.
Power of leg muscles | 2.5 hours after inclusion in study
  Peak power measured by countermovement jump performed on a force plate. Reported in N/kg
Arterial stiffness | 0.5 hours after inclusion in study
  Meausred by an noninvasive vascular screening system. Reported as brachial-ankle pulse wave velocity (baPWV).
Endothelial function | 1 hours after inclusion in study
  Meausred as flow mediated dilation (FMD) by ultrasound reported as %.
Left ventricular ejection fraction | 1 hour after inclusion in study
  Meausred by echocardiography reported as %.
Carotid-intima-media thickness | 1 hour after inclusion in study
  Carotid intima-media thickness (mm) is measured by 2D ultrasound instrument.
Retinal arterial and venous diameters | 7-30 days after inclusion in study
  Measured by static retinal vessel analysis. Diameters will be averaged to central retinal arteriolar and venular equivalents (CRAE and CRVE) and the arteriolar-to-venular diameter ratio will be calculated from the CRAE and CRVE.
Retinal endothelial function | 7-30 days after inclusion in study
  Measured by dynamic retinal vessel analysis reported as %.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Sport, Exercise and Health, Section Sports and Exercise Medicine, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwendinger F, Knaier R, Wagner J, Infanger D, Lichtenstein E, Hinrichs T, Rowlands A, Schmidt-Trucksass A. Relative and absolute intensity accelerometer metrics decipher the effects of age, sex, and occupation on physical activity. BMC Public Health. 2025 Mar 6;25(1):885. doi: 10.1186/s12889-025-21800-w. PMID 40050804
- [Derived] Prechtl L, Carrard J, Gallart-Ayala H, Borreggine R, Teav T, Konigstein K, Wagner J, Knaier R, Infanger D, Streese L, Hinrichs T, Hanssen H, Ivanisevic J, Schmidt-Trucksass A. Circulating amino acid signature features urea cycle alterations associated with coronary artery disease. Sci Rep. 2024 Oct 28;14(1):25848. doi: 10.1038/s41598-024-76835-7. PMID 39468229
- [Derived] Schwendinger F, Wagner J, Knaier R, Infanger D, Rowlands AV, Hinrichs T, Schmidt-Trucksass A. Accelerometer Metrics: Healthy Adult Reference Values, Associations with Cardiorespiratory Fitness, and Clinical Implications. Med Sci Sports Exerc. 2024 Feb 1;56(2):170-180. doi: 10.1249/MSS.0000000000003299. Epub 2023 Sep 12. PMID 37703330
- [Derived] Schwendinger F, Wagner J, Infanger D, Schmidt-Trucksass A, Knaier R. Methodological aspects for accelerometer-based assessment of physical activity in heart failure and health. BMC Med Res Methodol. 2021 Nov 14;21(1):251. doi: 10.1186/s12874-021-01350-6. PMID 34775952
- [Derived] Streese L, Vaes A, Infanger D, Roth R, Hanssen H. Quantification of Retinal Vessel Myogenic Constriction in Response to Blood Pressure Peaks: Implications for Flicker Light-Induced Dilatation. Front Physiol. 2021 Feb 18;12:608985. doi: 10.3389/fphys.2021.608985. eCollection 2021. PMID 33679432